CLINICAL TRIAL: NCT01734759
Title: Influence of Medication Palatability on Prescribing Habits of Pediatric Prescribers
Brief Title: Influence of Medication Taste on Pediatric Prescribers' Prescribing Habits
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bernard Lee, Principle Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-005823
Record Dates: First submitted 2012-11-17; First posted 2012-11-28 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: medication palatability; medication taste

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taste Test (Experimental)
  Interventions: Drug: Taste Test

INTERVENTIONS:
Drug: Taste Test — Before the taste test each participant will fill out an informed consent form and an enrollment survey. Each participant will receive 0.5 mL of each study medication in the taste test. During the taste test each medication in a class will be labeled with a color name so as to prevent any bias from preconceived taste perception. They will record their perception of the medications taste on a visual analog scale (VAS). An anaphlyaxis kit will be on hand in case of emergencies. Between samples participants will cleanse their palate with a saltine cracker and 30 mL of water. 5 different classes of medications will be tested.
  Medications to be sampled and the corresponding dose of the test dose are:
  * Cephalosporins: cefdinir 12.5 mg, cefixime 10 mg
  * Penicillins: penicillin VK 12.5 mg, amoxicillin 12.5 mg
  * Analgesic/antipyretics: acetaminophen 16 mg, ibuprofen 10 mg
  * Steroids: prednisolone 1.5 mg, prednisone 0.5 mg
  * H2 receptor blockers: famotidine 4 mg, ranitidine 7.5 mg

SUMMARY:
The purpose of this study is to see if a medication taste test influences the prescribing habits of pediatric prescribers at Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria:

* subjects possess prescriptive authority (e.g. MD, nurse practitioner, physician's assistant, medication therapy management pharmacists)
* subjects have prescribed at least one of the study medications from one of the medication classes to pediatric patients at an outpatient clinic in the three months preceding the study

Exclusion Criteria:

* subjects do not prescribe any of the tested medications
* subject has an allergy to all of the study medications
* subject is pregnant or breastfeeding
* subject has a medical condition that prevents them from being involved in the taste test

Participants are advised to be within or accessible to the Rochester, MN area during study recruitment and accessible afterwards via mail, email or fax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Taste scores on the visual analog scale | Change from baseline in taste scores at 3 months
  Medication taste scores on the visual analog scale before and after a medication tasting will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Lee, PharmD, RPh, Principal Investigator — Mayo Clinic; Ole J Olson, Pharm.D., BCPS, Principal Investigator — Mayo Clinic; Michelle J LoTurco, Pharm.D., Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States